CLINICAL TRIAL: NCT01369004
Title: The Use of Weight Tracking Technology to Promote Weight Loss Among Overweight Adults
Brief Title: The WEIGH Study: Weighing to Improve and Gain Health
Acronym: WEIGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-2013
Record Dates: First submitted 2011-06-02; First posted 2011-06-08 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2012-09

CONDITIONS: Overweight and Obesity
Keywords: self-weighing; self-monitoring; weight loss; obesity
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily self-weighing + feedback/lessons (Experimental): Participants will be instructed to weigh daily and they will receive a smart scale for daily monitoring of weighing via the website bodytrace.com. They will also receive weekly emailed lessons with content related to behavioral weight control (e.g., How to control portion sizes, How to develop an exercise routine) as well as weekly emailed feedback from a registered dietitian on their daily weighing and weight loss progress.
  Interventions: Behavioral: Daily Self-weighing + weekly feedback+ weekly lessons
- Delayed Intervention Control Group (No Intervention): Participants will receive the same components of the experimental group with the exception of the weekly feedback after the 6-month study period is complete.

INTERVENTIONS:
Behavioral: Daily Self-weighing + weekly feedback+ weekly lessons — Daily self-weighing as a form of self-monitoring of body weight using a smart scale that sends their weights directly to a website (www.bodytrace.com) via the cellular network. They will be able to review weight trends overtime on this website via a graph showing both changes in weight and BMI. They will also receive weekly emailed feedback on their weight loss progress and compliance to the daily self-weighing prescription from a registered dietitian, as well as weekly emailed lessons with content related to behavioral weight control (e.g, how to control portion sizes, how to develop and exercise routine).
  Other Names: Daily Self-weighing Intervention
  Arms: Daily self-weighing + feedback/lessons

SUMMARY:
The purpose of this research project is to assess the efficacy of a weight loss intervention for chronic disease prevention that focuses on daily self-weighing as the primary self-monitoring strategy compared to a delayed-intervention control group. While daily self-weighing has been shown to be effective for weight loss in observational research, there is limited experimental evidence testing this association and most is derived from intensive interventions that may overshadow the effects of self-weighing. To mitigate this, the investigators will examine whether daily self-weighing is effective for weight loss under self-directed conditions using a randomized-controlled design.

The investigators will conduct a 6-month randomized trial in 88 overweight and obese adults to compare a daily self-weighing intervention to a delayed-intervention control group. Changes in weight, diet and physical activity, and psychosocial measures will be examined.

Main Study Hypothesis: Participants in the group randomized to receive the daily self-weighing intervention will have greater percent weight loss at 6 months compared to those in the delayed control group.

Secondary Hypothesis: Participants in the group receiving the daily self-weighing intervention will report greater engagement in diet and physical activity behaviors that produce caloric deficits, greater self-efficacy and motivation, and no differences in body satisfaction, disordered eating, or depressive symptoms compared to those in the control group.

DETAILED DESCRIPTION:
Obesity continues to be a challenging public health problem. Despite producing large reductions in weight, weight loss interventions require a significant amount of effort because of the detailed self-monitoring of dietary intake and exercise habits that is involved. Consequently, this behavior is difficult to sustain and weight regain occurs. Interventions focused on enhancing simple strategies for self-monitoring may be just as effective and provide more lasting effects.

One of the simplest forms of self-monitoring is self-weighing. Self-weighing is an important tool for regulation of body weight as it provides proximal feedback on how eating and exercise behaviors are impacting weight, and allows individuals to make adjustments to these behaviors to affect energy balance. Observational research indicates that daily self-weighing is associated with greater weight loss as compared to less frequent self-weighing. However, there is limited experimental evidence testing this association and most is derived from intensive interventions that may overshadow the effects of self-weighing. To mitigate this, the investigators will examine whether daily self-weighing is effective under self-directed conditions with minimal contact. The results of this proposal will provide evidence about the efficacy of daily self-weighing on weight loss using a randomized controlled design. Most assessments of self-weighing are measured via self-report, which introduces measurement error. This proposal will improve on this by using an objective measure of self-weighing with a scale that can store and transmit weight data.

Given that self-weighing does not impact weight loss directly but rather via changes in diet and physical activity behaviors, a full understanding of the mechanisms explaining this relationship is necessary. Furthermore, despite evidence indicating that more frequent self-weighing has no adverse psychological effects in adults participating in weight control interventions, there remains debate as to the negative psychological consequences of this behavior. Therefore, it would be informative to test for any adverse effects between treatment groups to further add to the evidence surrounding this debate.

The objective of the WEIGH Study (Weighing to Improve and Gain Health) is to test the efficacy of a self-directed intervention focused on daily self-weighing as the main self-monitoring strategy on weight loss at 6 months compared to a delayed-intervention control group. This will be tested using a 2-group randomized control design. Participants will be randomly assigned to either: [1] Daily Self-weighing Intervention Group or [2] Delayed-Intervention control group. The daily self-weighing intervention group will receive access to a "smart scale" for daily self-weighing and viewing of weight trends over time, and receive weekly emails with tailored messages reinforcing self-weighing and other behaviors associated with reaching weight loss goals. This group will also receive weekly lessons with basic information for weight loss and strategies on how to use the scale to maximize weight loss. The control group will be given the "smart scale" and be told to weigh as often as they normally do, with the goal of observing natural weighing frequency trends in this group. After the end of the 6-month study, they will receive a 3-month modified version of the daily self-weighing intervention, which will include weekly emails, prescription for daily self-weighing, and weight monitoring via the smart scale website. Detailed descriptions of these components are outlined below.

Recruitment and Informed Consent Participants will first undergo screening at www.uncweightresearch.org via Qualtrics or call the study center to complete the screening questionnaire over the phone. For those filling out the questionnaire online, they are still required to call the study center to complete the screening questionnaire, as sensitive medical-related questions are more appropriate to ask over the phone.

Once they are considered eligible, participants will be invited to an orientation session where they can hear more about the program and ask any questions before deciding whether or not to participate. For those who want to participate, the study PI and/or other study personnel listed on this application will explain the consent form and ask the participant to read the form. Once the participant has finished reading the form, the study personnel member will ask the participant if he/she has any questions. Then both parties will sign the questionnaire and the participant will receive a copy of the consent form.

Randomization Consented individuals will be provided with a Qualtrics link to complete baseline questionnaire measures. A computer algorithm will randomly assign them to one of the two study groups. Baseline anthropometrics will be measured at the kick-off session where randomization will be revealed to all participants. At both the 3 and 6-month assessments, the enrolled patients will repeat all baseline measures, with the exception of demographic characteristics. At 9 months, participants in both groups will be asked to stop on their smart scale to provide a final weight measurement and the control group will complete 1 final questionnaire. Following randomization, participants will either receive the components outlined below for the intervention group or for the delayed-intervention control group.

Detailed Descriptions of the Intervention Components Kick-off Group Meeting Initially, individuals will attend a group kick-off meeting where they will receive scales (see below) and other materials for getting started. This meeting will also emphasize the objective of the study, which is to examine the effect of a self-directed approach for weight loss emphasizing daily self-weighing. The kick-off session will provide participants will a start-up guide for how to use the scale as well as access to the study website (www.bodytrace.com) for viewing of weight trends overtime. The session will focus on the benefits of daily self-weighing for weight loss, addressing certain myths regarding daily self-weighing and emphasizing the use of the scale as a barometer for progress with diet and physical activity behaviors. In addition, this session will also provide a brief overview of "Weight Loss 101" through a discussion focused on calorie balance, as it outlined in the Diabetes Prevention Program materials.

Smart Scales Participants in the intervention group will be instructed to weigh themselves daily using "smart" scales. These scales send weight data directly to a website (www.bodytrace.com) via the wireless cellular network. Participants will be able to view their weight on the scale and can also utilize the website to view weight trends overtime. Participants will be loaned these scales, and will be told in the consent form that they will be be able to keep the smart scale upon completion of all study assessment visits. Participants will be told that if they do not complete the assessment visits, they will be asked to return to the UNC Weight Research Program.

Intervention Weekly Emails All intervention participants will receive weekly emails that include basic skills training materials about weight control, and tailored feedback based on rate of weight loss and daily self-weighing frequency. The skills training materials will include instructional lessons about topics such as portion control, label reading, restaurant eating, structured exercise, and lifestyle activity, and behavioral topics such as problem solving, stimulus control and relapse prevention. The behavioral topics are based on the evidence based Diabetes Prevention Program. This program has been used in various research studies, including those conducted at the UNC Weight Research Program. Additionally, the investigators will reinforce self-weighing through behavioral weight control topics to enhance self-regulation.

The emails will begin with a tailored feedback message about daily self-weighing frequency and a message to reinforce daily self-weighing to help participants respond effectively to weight changes by learning how to utilize their scale to make adjustments to diet and physical activity behaviors in order to produce caloric deficits. An algorithm based on self-weighing frequency compliance will determine which feedback message they receive

Diet and Physical Activity Level Suggestions Participants in the intervention group will also receive examples of meal plans for each of the calorie levels associated with weight loss (e.g., 1200-1800 calories per day) and be given suggestions for which meal plan to follow based on baseline weight, Furthermore, all participants will be provided with a physical activity goal of 150-250 minutes per week of exercise similar to brisk walking, as this level is shown to be associated with weight loss. They will be encouraged to begin with 10 minutes of walking each day and to add 5 minutes per day each week until they reach the 150-200 minutes. For example, Week 1 walk 10 minutes x 5 days (50 minutes), Week 2 walk 15 minutes x 5 days (75 minutes), Week 3 walk 20 minutes x 5 days (100 minutes), etc.

Delayed-Intervention Control Group The delayed-intervention control group will receive a kick-off session where they will be told that the study is testing a self-directed approach to weight loss focusing on careful tracking of weight, and that they will receive a modified version of the intervention after the 6-month period is complete. They will also be provided with the "smart scales" but not website access (bodytrace.com), and be told to use them as they normally would, so that the investigators could get a sense of their normal weighing habits. They will be told that the investigators will be able to view their weighing frequency on the bodytrace.com website. They will receive a modified version of the intervention for 3 months, which will include the same components as the intervention group with the exception of the weekly feedback emails. After 3 months, the investigators will call and/or email participants to ask them to step on the scale and provide a final weight and complete 1 final questionnaire on process measures.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-60 years old
* Have a BMI between 25-40 kg/m^2 and weigh no more than 310 lbs.
* Live in the Chapel Hill/Durham/Raleigh, NC area
* Be able to attend data collection visits at baseline, 3-months, and 6-months at the UNC Weight Research Program Center
* Have access to the Internet and a computer for daily tracking of weight
* Be willing to be randomized to either group

Exclusion Criteria:

* History of psychiatric diseases (bipolar disorder, schizophrenia, hospitalization for depression within the past year), drug or alcohol dependency, or uncontrolled thyroid conditions
* History of major health conditions, such as heart disease, diabetes, and past incidence of stroke, cancer diagnosis (non-skin) within the past 5 years
* No physician consent for participation if currently on blood pressure medications, have issues with dizziness, or have bone or joint issues.
* Currently pregnant, anticipating on becoming pregnant in the next 9 months, or currently breastfeeding
* History of eating disorder or currently seeking treatment for an eating disorder.
* Current participation in a structured weight loss program,or taking weight loss medications
* Current participation in a weight control study within the past 6 months
* Current participation in another research study that might affect study hypotheses
* Have lost 5% of their body weight and kept it off within the past 6 months
* History of surgery for weight loss
* Plans to be out of the area for an extensive amount of time without Internet access or move out of the area within the next 9 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Percent Weight Loss | 6 months
  The primary outcome is percent weight loss at 6 months. Weight will be collected at baseline, 3, and 6 months at the UNC Weight Research Program Center and measured to the nearest 0.2 lbs using a digital Tanita scale that will be calibrated routinely. Participants will weigh-in wearing light clothes and no shoes

SECONDARY OUTCOMES:
Changes in Caloric Intake | 6 months
  Caloric intake will be assessed at baseline, 3 and 6 months using the online Automated Self-Administered 24-hour recall tool created by the National Cancer Institute.
Changes in Energy Expenditure from Exercise | 6 months
  Energy expenditure from exercise will be assessed at baseline, 3, and 6 months via the Paffenbarger Exercise Habits Questionnaire.
Changes in Self-efficacy for Eating Behaviors | 6 months
  We will assess self-efficacy for eating behaviors related to weight control at baseline, 3 and 6 months using the Weight Efficacy Lifestyle Questionnaire.
Changes in self-efficacy for exercise behaviors | 6 months
  We will assess self-efficacy for exercise behaviors at baseline, 3 months, and 6 months using the Sallis Self-efficacy for Exercise Behaviors Questionnaire.
Changes in Weight Control Strategies (diet and exercise) | 6 months
  At baseline, 3months, and 6 months, we will assess behavioral strategies (both diet and exercise) associated with successful weight control using the Eating Behavior Inventory and the Weight Management Strategies Questionnaire. These strategies have been shown to be associated with greater weight loss in other weight control trials.
Changes in Motivation | 6 months
  We will assess autonomous and controlled motivation at baseline, 3 months, and 6 months using the Treatment Self-Regulation Questionnaire.
Changes in Dietary Hunger, Restraint, and Disinhibition | 6 months
  We will assess dietary hunger, restraint, and disinhibition at baseline, 3 months, and 6 months using the Three Factor Eating Questionnaire.
Changes in Binge Eating symptoms | 6 months
  The Questionnaire on Eating and Weight Patterns-Revised will be administered at baseline, 3 months, and 6 months to assess changes in behaviors related to binge eating and bulimia.
Changes in depressive symptoms | 6 months
  The Center for Epidemiologic Studies Depression Scale will be used to assess depressive symptoms at baseline, 3 months, and 6 months.
Changes in Body Shape Concerns | 6 months
  The Body Shape Questionnaire will be used to assess changes in body shape concerns at baseline, 3 months, and 6 months.
Changes in cognitions related to disordered eating | 6 months
  Disordered eating cognitions, patterns, and behaviors will be assessed using a brief version of the Mizes Anorectic Cognitions Questionnaire (BMAC-Q) at baseline, 3 months, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dori M Steinberg, PhD, MS, RD, Principal Investigator — University of North Carolina, Chapel Hill; Deborah Tate, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- UNC Weight Research Program, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Steinberg DM, Tate DF, Bennett GG, Ennett S, Samuel-Hodge C, Ward DS. Daily self-weighing and adverse psychological outcomes: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):24-9. doi: 10.1016/j.amepre.2013.08.006. PMID 24355668